CLINICAL TRIAL: NCT03917368
Title: Validation of a Novel Non-invasive Technique Based on Real-time Ultrasound B-mode to Assess the Jugular Venous Pulse
Brief Title: Ultrasound Evaluation of the Jugular Venous Pulse (US-JVP)
Acronym: US-JVP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: S. Anna Hospital (Other)
Responsible Party: Principal Investigator, Paolo Zamboni, Full Professor, Director Vascular Diseases Center, University of Ferrara, S. Anna Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RF-2013-02358029
Record Dates: First submitted 2019-03-19; First posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Emergencies; Cardiovascular Diseases; Neurovascular Disorders
Keywords: Jugular Venous Pulse; Central Venous Pressure; Ultrasounds; Validation Studies; Software Validation
MeSH Terms: conditions — Emergencies; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound scan of the internal jugular veins (Experimental): Hospitalised adult patients, requiring a scheduled central venous catheterisation and measurement of the central venous pressure as part of their usual care, will undergo a non-invasive ultrasound scan of the internal jugular veins (both side of the neck) synchronized with an ECG trace, to assess the jugular venous pulse. This procedure will be performed once throughout the study.
  Interventions: Other: Ultrasound scan of the internal jugular veins

INTERVENTIONS:
Other: Ultrasound scan of the internal jugular veins — Participants, lying at their hospital bed, will maintain their head in a fixed position on the longitudinal axis, while an operator gently places a linear probe L12-RS (7.5-11 MHz), smeared with gel, on one side of the neck, at the middle level. A 15-sec video clip of the ultrasound images will be recorded. This procedure will be repeated on the other side of the neck. In addition, three electrodes will be placed on participants' chests and connected to the ultrasound system for simultaneously measuring the ECG signal.

SUMMARY:
The jugular venous pulse (JVP) reflects changes in the right atrial pressure and its evaluation can be useful in managing many emergency conditions for guiding the fluid administration as well as in the diagnosis and/or prognosis of many heart and lung diseases. The present study aims: i) To validate a novel ultrasonographic (US) technique for obtaining the JVP from a high-resolution B-mode sonograms sequence, recording the changes of the cross-sectional area (CSA) of the internal jugular veins (IJV) over the cardiac cycle; ii) To develop physical and mathematical models capable of providing an indirect estimate of central venous pressure (CVP) from the changes in IJV-CSA acquired through the US investigation, and iii) To test the transferability of the novel US-JVP technique in a clinical setting.

DETAILED DESCRIPTION:
The study will be articulated in different phases, encompassing data collection, development of physical and mathematical models, statistical evaluations, and software implementation. The clinical experimental phase of the study (data collection) will involve hospitalized adult patients requiring a scheduled central venous catheterization and measurement of the CVP as part of their usual care. The latter will be used as the gold standard measure of CVP for the subsequent data processing and analysis. A small sample of healthy adult volunteers will also be recruited only for the non-invasive US evaluation of the JVP. The validation processes will include assessment of the diagnostic power of the US-JVP estimated CVP values and US-JVP waveforms, including evaluation of sensibility, specificity, predictive positive and negative values, accuracy and precision.

ELIGIBILITY:
Inclusion criteria:

* Adult (age ≥18 years) hospitalized patients, spontaneous breathing, requiring a scheduled central venous catheterization and measurement of the central venous pressure as part of their usual care;
* Capacity to give informed consent.

Exclusion criteria:

* Central venous catheterization via the internal jugular venous access

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-09-16 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Jugular venous pulse by ultrasound | 1 day
  Internal jugular vein cross sectional area variations in cm2 over a cardiac cycle obtained from a high-resolution B-mode sonograms sequence.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Zamboni, Prof, Principal Investigator — University Hospital of Ferrara, Italy
Locations (1):
- University Hospital of Ferrara, Ferrara, Italy